CLINICAL TRIAL: NCT04258748
Title: Effect of Motivational Interviewing and Game Based Education on Oral Hygiene Behavior of Preschool Children in Beheira Governorate, Egypt
Brief Title: Effect of Motivational Interviewing and Game Based Education on Oral Hygiene Behavior of Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Instructor of Dental Public Health and Statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MI and game based education
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Motivation
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivational Interviewing (MI) (Experimental)
  Interventions: Behavioral: Motivational Interviewing (MI)
- Gaming and MI (Experimental)
  Interventions: Behavioral: Gaming and MI
- Conventional dental health education (Active Comparator)
  Interventions: Behavioral: Conventional dental health education

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) — In each of the four MI counseling sessions that were delivered, the researcher approached mothers in small groups of 5 via three phases, in 15-30 minutes, to establish rapport/ alliance in the first phase, to identify health needs in the second phase and finally to reinforce dental needs in the third phase.
  Arms: Motivational Interviewing (MI)
Behavioral: Gaming and MI — In each of the four MI counseling sessions, the researcher approached mothers via three phases, in 15-30 minutes, to establish rapport/ alliance, to identify and finally reinforce dental needs in the same pattern as MI group. In addition, the children were engaged in 'Happy Teeth, Healthy Kids' which is an android tablet game that was included in the MI session scheduled for the mothers. Children were told to follow correct steps of brushing in order to obtain happy bright teeth. This helped the children realize that brushing teeth will give them a bright smile.
  Arms: Gaming and MI
Behavioral: Conventional dental health education — It was delivered through a 15-minutes oral health session given to mothers of preschoolers. Mothers were given brief information about causes of dental caries and role of plaque, toothbrush size, diet / frequency of sweet snacks, brushing technique, toothpaste and fluoride use as well as regular dental visits. Participants were then shown a short educational video about prevention of dental caries among children coupled with oral hygiene instructions. At the end of the session, participants were given a leaflet reinforcing the information to take home.
  Arms: Conventional dental health education

SUMMARY:
The purpose of this study was to evaluate the effectiveness of motivational interviewing as well as games in changing oral health behaviors among preschool children.

DETAILED DESCRIPTION:
The participating children, in this randomized controlled clinical trial, were recruited from the governmental preschools available within Edko administration of Beheira governorate, Egypt. A cluster random sampling strategy was used so that the contributors, after fulfilling eligibility criteria, mother/child dyads (pairs) in each nursery were subsequently assigned to the first test group (motivational interviewing MI), the second test group (motivational interviewing MI+ gaming) or the control group (conventional dental health education CE). The children were randomly assigned to the three study groups in the allocation ratio 1:1:1 using random allocation software in blocks of five. The schools' randomization sequence were written on identical sheets of paper and folded inside opaque envelopes that were sealed to be open at the time of intervention implementation.

The three interventions were the conventional dental health education (CE) which were delivered through a 15-minute oral health session given to mothers of preschoolers in the control group whereas in the test groups Motivational Interviewing (MI) for mothers and Games for children were carried out via specific phases.

ELIGIBILITY:
Inclusion Criteria:

* Children having unfavorable oral health behavior (reporting a maximum tooth brushing frequency of 1-2 times/ week).
* The child's mother agreed to join the study so that parent/child can be recruited as pairs/dyads.
* Children enrolled in one of the nurseries selected

Exclusion Criteria:

* Children having a history of serious medical condition or special care needs
* Using any type of removable appliances such as space maintainer or tongue guard.
* Children whose mothers refused to give consent to participate in the study.
* Illiterate mothers who were not able to understand the oral health materials and instructions.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-01-05 (Actual)

PRIMARY OUTCOMES:
Rate of dental plaque accumulation | baseline
  It was assesed using modified OHI-S.The presence of plaque was verified on the buccal surface of 6 index teeth: the upper right second deciduous molar (tooth 55), the upper right central deciduous incisor (tooth 51), the upper left second deciduous molar (tooth 65), the lower right second deciduous molar (tooth 85), the lower left central deciduous incisor (tooth 71), and the lower left second deciduous molar (tooth 75). According to the OHI-S, dental plaque is defined as a soft organic material loosely adhering to the tooth surface. The tooth surface covered by plaque was estimated by visual examination according to the following criteria: 0 =no plaque present; 1 = plaque covering no more than 1/3 of the surface in question; 2 = plaque covering more than 1/3, but no more than 2/3 of the surface; 3= plaque covering more than 2/3 of the surface; 9 = tooth excluded, no information.
Rate of dental plaque accumulation | 6 months
  It was assesed using modified OHI-S.The presence of plaque was verified on the buccal surface of 6 index teeth: the upper right second deciduous molar (tooth 55), the upper right central deciduous incisor (tooth 51), the upper left second deciduous molar (tooth 65), the lower right second deciduous molar (tooth 85), the lower left central deciduous incisor (tooth 71), and the lower left second deciduous molar (tooth 75). According to the OHI-S, dental plaque is defined as a soft organic material loosely adhering to the tooth surface. The tooth surface covered by plaque was estimated by visual examination according to the following criteria: 0 =no plaque present; 1 = plaque covering no more than 1/3 of the surface in question; 2 = plaque covering more than 1/3, but no more than 2/3 of the surface; 3= plaque covering more than 2/3 of the surface; 9 = tooth excluded, no information.

CONTACTS AND LOCATIONS:
Overall Officials: Amani Nomair, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Maha Hamza, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Wafaa Essameldin, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Governmental nurseries within Edko administration, Beheira, Egypt